CLINICAL TRIAL: NCT00499161
Title: Effect of Patient-Centered Care (PCC) on Patient Satisfaction at Hospital Discharge
Acronym: PCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Debra M. Wolf, PhD, MSN, RN, University of PIttsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PRO07030017
Record Dates: First submitted 2007-07-09; First posted 2007-07-11 (Estimated); Last update posted 2008-02-18 (Estimated); Status verified 2008-02

CONDITIONS: Patient Centered Care
Keywords: Individualized care; Relationship based care; Negotiated care; Patient focused care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Control group received usual care
- 2 (Experimental): Received intervention New model of nursing care
  Interventions: Behavioral: New model of nursing care

INTERVENTIONS:
Behavioral: New model of nursing care
  Arms: 2

SUMMARY:
The purpose of this randomized clinical trial is to examine the effect of Patient-Centered Care (PCC) on a patient's level of satisfaction on discharge from an acute healthcare setting. Findings from this study will assist in determining if PCC, administered by nurses, should be instituted hospital wide.

SPECIFIC AIMS:

1. To examine the effect of Patient-Centered Care on patient satisfaction.
2. To examine the effect of Patient-Centered Care on the quality of patient care.
3. To examine the effect of patient's perception of nursing care on patient satisfaction.

DETAILED DESCRIPTION:
Patient-Centered Care (PCC), also known as individualized patient care or negotiated care, focuses on the patient's right to have his/her values and beliefs respected as an individual.This respect is viewed as part of a commitment to build a deep understanding of the patient as a thinking and feeling individual with the ability to change and develop. A person-centered model of care requires a nurse to work with an individual's beliefs, values, wants, needs and desires.This adaptation to a patient's personal needs requires the nurse to be flexible, respectful, and reciprocal when providing patient care. If the patient's expectations are not appropriate to the type of care needed to heal or if the patient refuses or denies a specific type of treatment that is known as influencing ones quality of care, the nurse must negotiate with the patient. Negotiation incorporates education, which is believed to increase the patient's level of understanding. In addition, negotiation allows the nurse and patient to define a level of treatment that is specific to the patient's needs but still seen as a quality indicator.

The Institute of Medicine (IOM) has listed PCC as one of six national quality aims for improvement. The IOM's vision is that all health professionals will be educated to provide and deliver PCC as part of an interdisciplinary team. In 2001, the IOM report "Crossing the Quality Chasm: A New Health System for the 21st Century" recommends a mixture of approaches to achieve their vision . These approaches include an appropriate training environment, research, public reporting and leadership. At present, there is little evidence to support the critical role nurse clinicians' play in providing PCC and satisfying patient's needs.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Admitted to the service of Dr.RQ and scheduled for bariatric bypass surgery
* Expected length of hospital stay ≥ 2 days.

Exclusion Criteria:

* Any prior admission to the study unit
* Bariatric surgery performed by a surgeon other than Dr.RQ
* Scheduled to have a LAP Band procedure, as this procedure has a different postoperative course.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-04; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Measure level of overall satisfaction | day of discharge

SECONDARY OUTCOMES:
Measure level of quality of care - 1)Length of stay, 2)infection, 3)falls | day of discharge and 7 days post discharge
measure satisfaction with nursing care | day of discharge
measure level of quality care (unplanned adverse events) | approximately 30 days post discharge

CONTACTS AND LOCATIONS:
Overall Officials: Debra M Wolf, MSN, Principal Investigator — University of Pittsburh, School of Nursing & UPMC St. Margaret; Lisa Lehman, BSN, Principal Investigator — University of Pittsburgh; Robert Quinlin, MD, Principal Investigator — University of Pittsburgh; Jodi Miller, BSN, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC St. Margaret, Pittsburgh, Pennsylvania, United States